CLINICAL TRIAL: NCT01076790
Title: The Effect of Dexmedetomidine on Reactivity to Noxious Stimuli During Propofol-remifentanil Anaesthesia and Surgery
Brief Title: Dexmedetomidine-propofol-remifentanil Anaesthesia and Reactivity to Noxious Stimuli
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arvi Yli-Hankala (Other)
Responsible Party: Sponsor-Investigator, Arvi Yli-Hankala, Professor, Tampere University Hospital
Organization: Tampere University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Kotoe_01; 2009-014619-11 (EudraCT Number)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Anaesthesia
Keywords: Nociception; Dexmedetomidine; Electroencephalogram; Electromyogram; Entropy Index; Bispectral Index; Electrocardiogram; Plethysmogram; Heart; Heart rate; Heart rate variability; Surgery
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexmedetomidine (Active Comparator): Analgo-sedative, adjuvant of propofol anesthesia
  Interventions: Drug: Dexmedetomidine; Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion 1 mcg/kg in 10 minutes; thereafter 0.7 mcg/kg/h until 30 minutes has elapsed from skin incision.
  Other Names: Precedex. CAS 113775476.
Drug: Saline — Saline infusion 1 mcg/kg in 10 minutes; thereafter 0.7 mcg/kg/h until 30 minutes has elapsed from skin incision.

SUMMARY:
Dexmedetomidine acts at central nervous system (specifically: at locus caeruleus), providing sedative and analgesic effects. It is widely used in intensive care. Surgery-related interventions elicit arousal ('nociceptive') reactions. The effects of dexmedetomidine on the neurophysiological signs of arousal are studied in surgical patients. Brain waves, electrocardiogram, Entropy Index, Bispectral Index, and fingertip pulse waves are recorded and analyzed later on. The course of anaesthesia and surgery are recorded.

DETAILED DESCRIPTION:
The patients are randomized to receive either dexmedetomidine or saline infusion before and during anaesthesia (dexmedetomidine 0.1 mcg/kg within 10 minutes, thereafter 0.7 mcg/kg/h until 30 min after skin incision).

Multi-channel EEG, Entropy, BIS, multi-channel EMG, ECG, and plethysmogram are recorded on computer. Anaesthesia and surgery associated events are annotated on computer.

Time points of endotracheal intubation, skin incision, and course of surgery well be analyzed in detail. Additionally, tetanic stimulus of ulnar nerve will be applied for each patient, and reactions to the stimulus will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* males or females giving informed consent
* age range 18-70 years
* elective surgery: laparoscopy, laparotomy, breast surgery
* general anaesthesia
* ASA classification 1 or 2

Exclusion Criteria:

* pregnancy
* body mass index 30.1 or more
* diseases affecting CNS, autonomic nervous system, heart, heart rate, or circulation
* chronic use of drugs affecting CNS, autonomic nervous system, heart, heart rate, or circulation; except antihypertensives, which are acceptable in this study
* chronic use of clonidine
* serious psychiatric disease or condition
* overuse of alcohol
* use of illicit drugs
* unability of understand, read or use Finnish language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Physiological reaction to noxious stimulus | 30 minutes
  Nociception-associated changes in EEG, EMG, Entropy Index values, BIS Index values, morphology of plethysmogram or ECG, heart rate, or hear rate variability.

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Yli-Hankala, MD, Study Chair — Tampere University Hospital; Arvi Yli-Hankala, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland